CLINICAL TRIAL: NCT02510274
Title: A Phase 1, Single and Multiple Dosing Study to Evaluate Pharmacokinetics and Pharmacodynamics of ASP3325 in Patients With Chronic Kidney Disease and Hyperphosphatemia Undergoing Hemodialysis
Brief Title: Single and Multiple Dosing Study in Hemodialysis Patients With Hyperphosphatemia in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3325-CL-0003
Record Dates: First submitted 2015-07-08; First posted 2015-07-29 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease; Hyperphosphatemia Undergoing Hemodialysis
Keywords: Hyperphosphatemia; ASP3325; Chronic Kidney Disease; pharmacodynamics; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — ASP3325

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part1, ASP3325 Tablet A (Experimental): ASP3325 tablets A will be orally administered with 150 mL of water in fasting condition on non-dialysis day in Day 1
  Interventions: Drug: ASP3325
- Part2, ASP3325 Tablet B group 1 (Experimental): ASP3325 tablets B will be orally administered t.i.d. 30 minutes before each meal for 2 weeks
  Interventions: Drug: ASP3325
- Part2, ASP3325 Tablet B group 2 (Experimental): ASP3325 tablets B will be orally administered t.i.d. 30 minutes just after each meal for 2 weeks
  Interventions: Drug: ASP3325

INTERVENTIONS:
Drug: ASP3325 — oral

SUMMARY:
The objective of this study is to assess PK, safety and tolerability of a single oral dose of ASP3325 and to assess PD, PK and safety of repeated oral doses of ASP3325 administered t.i.d. before or just after each meal

DETAILED DESCRIPTION:
[Part 1] This part is an open-label, uncontrolled study to evaluate PK and safety with single dosing of ASP3325 in hemodialysis patients. After washout period of therapeutic medication for hyperphosphatemia, six subjects will receive single oral administration of ASP3325 (Tablet A) on a non-dialysis day (Day 1).

[Part 2] This part is a 2-arm, open-label, uncontrolled study to evaluate PD, PK and safety with dosing ASP3325 Tablet B t.i.d. before or just after each meal.

Eligible subjects at screening will be entered into the washout period for stopping their phosphate-binding treatment. 20 subjects with serum inorganic phosphorus (Pi) level between ≥6.0 and <10.0 mg/dL during the washout period (washout period week 1 or washout period week 2) will be randomized to each treatment group and ASP3325 will be administered for 2 weeks until Day 14.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has received maintenance hemodialysis 3 times a week for at least 12 weeks (84 days) prior to the scheduled first day of the washout period.
* Subject who can receive morning dialysis from the start of the washout period to the end of follow-up period. (Part 2)
* Subject with pre-dialysis serum Pi level between ≥6.0 and <10.0 mg/dL and be confirmed increase in serum Pi of ≥1.5 mg/dL after the maximum dialysis interval at the washout period week 1 or 2. (Part 2)
* Subject who did not change the type or dose of any phosphate binder(s), any nutritional supplements or any other drugs with phosphorus reducing action for at least 4 weeks (28 days) prior to the scheduled first day of the washout period.
* Subject who did not receive calcimimetics (e.g., cinacalcet HCl) for at least 12 weeks (84 days) prior to the scheduled first day of the washout period.
* Subject taking native or active vitamin D (including vitamin D analogues), calcitonin agents or PTH agents must be on stable dose for at least 4 weeks (28 days) prior to the scheduled first day of the washout period.

Exclusion Criteria:

* Subject who has a history of severe gastrointestinal disorder, major gastrointestinal surgery, malabsorption considered influential on the absorption of the drug and nutrition in the gastrointestinal tract.
* Subject who has a history of parathyroid intervention (e.g., parathyroidectomy [PTx], percutaneous ethanol injection therapy [PEIT]).
* Subject whose dry weight loss >5% within 12 weeks (84 days) prior to the scheduled start day of the washout period.
* Confirmed serum intact PTH >1000 pg/mL at the start of the washout period (only applicable for Part 2).
* Subject whose last 3 measurement values at the separate day of pre-dialysis systolic/diastolic blood pressure before the scheduled start day of the washout period or during the washout period are all 180 mmHg or higher and 120 mmHg or higher.
* Subject who has severe congestive heart failure (i.e., NYHA cardiac function classification Class III or severer).
* Subject who experienced a myocardial infarction or major surgery excluding vascular access surgery within 12 weeks (84 days) prior to the informed consent signing.
* Subject who has any of liver function tests (ALT, AST, T-Bil) out of range as indicated below at the screening (Part 1) or during the washout period, or patients with a complication of serious hepatic disease (e.g., acute and active chronic hepatitis, liver cirrhosis). AST: >2×ULN, ALT: >2×ULN, T-Bil: >1.25×ULN
* Subject with history or complication of malignant tumor (considered eligible if recurrence has not been observed for at least 5 years).
* Subject with history of serious drug hypersensitivity, such as anaphylactic shock.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2014-11-04 (Actual); Study Completion 2014-11-04 (Actual)

PRIMARY OUTCOMES:
Safety assessed by adverse events: Part 1 | Up to Day 7
Safety assessed by adverse events: Part 2 | Up to Day 22
Safety assessed by vital signs: Part 1 | Up to Day 7
  Vital signs include body temperature, blood pressure and pulse rate)
Safety assessed by vital signs: Part 2 | Up to Day 22
  Vital signs include body temperature, blood pressure and pulse rate)
Safety assessed by clinical laboratory test: Part 1 | Up to Day 7
  Clinical laboratory tests include hematology and biochemistry
Safety assessed by clinical laboratory test: Part 2 | Up to Day 22
  Clinical laboratory tests include hematology and biochemistry
Safety assessed by 12-Lead ECG: Part 1 | Up to Day 7
  ECG: electrocardiogram
Safety assessed by 12-Lead ECG: Part 2 | Up to Day 22
  ECG: electrocardiogram

SECONDARY OUTCOMES:
Cmax of unchanged ASP3325 | Part 1 Before administration, Day 1, 2, 4, 5 and 7
  Cmax:maximum plasma concentration
tmax of unchanged ASP3325 | Part 1 Before administration, Day 1, 2, 4, 5 and 7
  tmax = time to reach maximum plasma concentration
AUClast of ASP3325 | Part 1 Before administration, Day 1, 2, 4, 5 and 7
  AUClast: Area under the Curve of plasma concentration during observation period in each observational day
AUCinf of ASP3325 | Part 1 Before administration, Day 1, 2, 4, 5 and 7
  AUCinf: Area under the Curve of plasma concentration
t1/2 of ASP3325 | Part 1 Before administration, Day 1, 2, 4, 5 and 7
  t1/2 = apparent terminal elimination half-life
Vz/F of ASP3325 | Part 1 Before administration, Day 1, 2, 4, 5 and 7
  Vz/F = apparent volume of distribution
CL/F of ASP3325 | Part 1 Before administration, Day 1, 2, 4, 5 and 7
  CL/F = oral clearance
Ctrough of ASP3325 | Part 2 Before administration, Day 3, 5, 8, 10, 12, 15 and 22
  Ctrough = observed trough concentration
Serum Pi of ASP3325 | Part 2 Day -21, -14, and -7 in washout period, Day 1, 8, 15 and 22
  Serum Pi: serum phosphate concentration before dialysis
Serum Calcium (adjusted for albumin) | Part 2 Day -21, -14, and -7 in washout period, Day 1, 8, 15 and 22
  Corrected value of Calcium (Ca) (mg/dL) = Observed value of Ca (mg/dL) + [4-albumin (g/dL)
Serum concentration of intact PTH before dialysis | Part 2 Day -21 in washout period, Day 1, 8, 15 and 22
  PTH = parathyroid hormone
Serum concentration of FGF23 | Part 2 Day -21 in washout period, Day 1, 8, 15 and 22
  FGF23 = fibroblast growth factor 23

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Site: 4, Aichi
  - Site: 5, Aichi
  - Site: 1, Ibaraki
  - Site: 2, Ibaraki
  - Site: 3, Shizuoka

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=273